CLINICAL TRIAL: NCT00287976
Title: Irinotecan Single-Drug Treatment For Children With Refractory or Recurrent Hepatoblastoma
Brief Title: Irinotecan in Treating Young Patients With Refractory or Recurrent Hepatoblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454758; CCLG-LT-2003-01; CCLG-IRINOTECAN; EU-20589
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Liver Cancer
Keywords: childhood hepatoblastoma; recurrent childhood liver cancer
MeSH Terms: conditions — Liver Neoplasms; Hepatoblastoma | interventions — Irinotecan

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well irinotecan works in treating young patients with refractory or recurrent hepatoblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the biological activity of irinotecan hydrochloride, when given on a prolonged schedule, in terms of response rate and rate of early progression, in young patients with refractory or recurrent hepatoblastoma.

Secondary

* Determine the duration of response in patients showing stable disease or an objective response (partial or complete response) to this drug.
* Determine the time to progression and overall survival of patients treated with this drug.
* Determine the rate of resectability in patients treated with this drug.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive irinotecan IV over 1 hour on days 1-5 and 8-12. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo evaluation for tumor resectability after courses 2, 3, or 4. Patients whose disease is considered resectable at any of these time points proceed to surgery.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatoblastoma

  * Refractory or recurrent disease

    * Failed prior first-line or second-line treatment
  * Metastatic disease allowed
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Elevated serum alpha-fetoprotein (AFP) allowed
* No hepatocellular carcinoma

PATIENT CHARACTERISTICS:

* Lansky performance status 50-100% in patients ≤ 10 years of age OR Karnofsky performance status 50-100% in patients > 10 years of age
* Life expectancy > 8 weeks
* Hemoglobin > 8 g/dL
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Serum bilirubin ≤ 2 times normal
* AST/ALT ≤ 2 times normal
* Serum creatinine ≤ 3 times normal
* Normal metabolic parameters (i.e., serum electrolytes, glucose, calcium, and phosphate)
* Not pregnant or nursing
* No severe uncontrolled infection or enterocolitis

PRIOR CONCURRENT THERAPY:

* Recovered from toxicity of prior therapy
* No chemotherapy within 3 weeks prior to study entry
* No prior irinotecan
* No other concurrent anticancer therapy

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-04; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Best overall response (complete response and partial response)

SECONDARY OUTCOMES:
Early progression
Death
Disease progression or recurrence
Surgical resection (complete or incomplete)

CONTACTS AND LOCATIONS:
Overall Officials: Jozsef Zsiros, MD, PhD, Study Chair — Emma Kinderziekenhuis; Laurence Brugieres, MD — Gustave Roussy, Cancer Campus, Grand Paris; Penelope Brock, MD, PhD — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (22):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- Emma Kinderziekenhuis, Amsterdam, Netherlands
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales